CLINICAL TRIAL: NCT06203366
Title: Effect of Vojta Therapy on Upper Extremity Function of Children With Cerebral
Brief Title: Effect of Vojta Therapy on Upper Extremity Function of Children With Cerebral Palsy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mahidol University (Other)
Collaborators: Srisangwan School (Unknown); SRI International (Industry); the royal patronage of crippled children (Unknown)
Responsible Party: Principal Investigator, Sivaporn Vongpipatana, Assistant Professor, Mahidol University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: MURA2023/780
Record Dates: First submitted 2023-11-30; First posted 2024-01-12 (Actual); Last update posted 2024-09-24 (Actual); Status verified 2024-09

CONDITIONS: Cerebral Palsy; Upper Extremity; Vojta Therapy
MeSH Terms: conditions — Cerebral Palsy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): * got the Vojta treatment 30 minutes/session, 3 times/week for 8 weeks
  * got the ADL and kinetic activities training 30 minutes, 3 times/week for 8 weeks
  Interventions: Procedure: Vojta therapy
- control group (No Intervention): - got the ADL and kinetic activities training 30 minutes, 3 times/week for 8 weeks

INTERVENTIONS:
Procedure: Vojta therapy — Vojta therapy is an old treatment method which was discovered by Professor Vaclav Vojta, a neurologist and pediatrician. It has been used to treat children with impair motor function in Thailand since 2011. Vojta therapy encourage the movement of children via positioning and stimulate the specified zone.
  Arms: Experimental group

SUMMARY:
The goal of this pilot study is to study the effect of Vojta therpy on upper extremity function in children with cerebral palsy. The main questions are:

* to study the effect of Vojta therapy on upper extremity function in children with cerebral palsy in terms of range of motion and function
* to study the effect of Vojta therapy on upper extremity function in children with cerebral palsy in terms of motion analysis while perform function

DETAILED DESCRIPTION:
Vojta therapy is an old treatment method which was discovered by Professor Vaclav Vojta, a neurologist and pediatrician. It has been used to treat children with impair motor function in Thailand since 2011. Vojta therapy encourage the movement of children via positioning and stimulate the specified zone.

ELIGIBILITY:
Inclusion Criteria:

* spastic diplegia (MACS II-III)
* can pick box and block test at least 1 block
* has good trunk stability while sitting
* can follow command
* participant and guardian consent to the study

Exclusion Criteria:

* no Vojta therapy in last 2 months
* no history of anti-spastic injection in last 6 months
* do not receive prednisolone nor adrenocorticotropic hormone (ACTH)
* cannot control seizure
* got the specific disease such as osteogenesis imperecta, cardiac disease
* Participant and guardians do not consent to the study.

Ages: 7 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 20 (Actual)
Dates: Start 2023-11-15 (Actual); Primary Completion 2024-08-30 (Actual); Study Completion 2024-08-30 (Actual)

PRIMARY OUTCOMES:
Box and block test | Baseline (before) and within 1 week after the final treatment
  the children have to pick the 1"*1" cube blocks from one side of the box to the other side in 1 minute

SECONDARY OUTCOMES:
active range of motion of upper extremity | Baseline (before) and within 1 week after the final treatment
  the children was asked to active move their shoulder, elbow and wrist for measurement
Nine hole peg test | Baseline (before) and within 1 week after the final treatment
  the children have to pick 9 pegs from the container to insert into the providing holes and record the time
3D motion analysis of upper extremity | Baseline (before) and within 1 week after the final treatment
  the markers were attached at back, sternum, both shoulders, elbows and wrists. Then, children were to forward rech the object on the table. The camera and mrakers will record and analyz the motion of both upper extremities. This measurement will be done only in children who was treated with Vojta therapy group only. This measurement will report in distance of maximum reaching, velocity and angle velocitym of shoulder, elbow, wrist with forearm pronation/supination. The other parameters are movement duration, peak velocity, time to peak velocity and trajectory straigthness.
Video recording | Baseline (before) and within 1 week after the final treatment
  The camera video will record the distance of maximum reaching in forward reaching and lateral reaching during the 3D kinematics evaluation in the gait lab of both upper extremities movement. This outcome was done in only the intervention group who received Vojta treatment.

OTHER OUTCOMES:
Kinect sensor | This outcome will be measured only in the intervention group. It will be measured immediately or not longer than 1 week after finish the intervention.
  The Kinect sensor evaluation of both upper extremities during playing computer game. Children will be asked to move their upper extremities according to game instructions: arm abduction/adduction, arm forward flexion/extension and elbow flexion/extension. During playing the computer game, there is a kinect sensor to detect motion of upper extremities and capture motion of movement in terms of range of motion, angle of movement in 3 dimensions and velocity of movements. while children playing game, there are recording of the movement via 3D motion analysis from gait lab. The parameters from Kinect sensor will be compared to the parameters which are recorded from the gait lab.

CONTACTS AND LOCATIONS:
Locations (1):
- Srisangwan School Foundation for the Welfare of the Crippled under Royal Patronage of Her Royal Highness the Princess Mother, Nonthaburi, Thailand

IPD SHARING:
Plan to Share IPD: Yes
For the study protocol and informed consent, they will be shared to all of the researchers. for the study protocol, SAP, ICF,CSR and analytic code, they will he shared to Chananchida Widchayasart and Parit Wongphaet after finishing data collection.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: after data collection

REFERENCES:
- [Background] Bax M, Goldstein M, Rosenbaum P, Leviton A, Paneth N, Dan B, Jacobsson B, Damiano D; Executive Committee for the Definition of Cerebral Palsy. Proposed definition and classification of cerebral palsy, April 2005. Dev Med Child Neurol. 2005 Aug;47(8):571-6. doi: 10.1017/s001216220500112x. PMID 16108461
- [Background] Sadowska M, Sarecka-Hujar B, Kopyta I. Cerebral Palsy: Current Opinions on Definition, Epidemiology, Risk Factors, Classification and Treatment Options. Neuropsychiatr Dis Treat. 2020 Jun 12;16:1505-1518. doi: 10.2147/NDT.S235165. eCollection 2020. PMID 32606703
- [Background] Prusmetikul S, Vongpipatana S, Woratanarat P, Tuntiyatorn P, Tamonsawatruk T. Correlation of range of motion and functional performance of upper extremities in children with cerebral palsy. J Med Assoc Thai 2018;101;Suppl.3
- [Background] Peeters LHC, de Groot IJM, Geurts ACH. Trunk involvement in performing upper extremity activities while seated in neurological patients with a flaccid trunk - A review. Gait Posture. 2018 May;62:46-55. doi: 10.1016/j.gaitpost.2018.02.028. Epub 2018 Mar 6. PMID 29524797
- [Background] Kara OK, Yardimci BN, Sahin S, Orhan C, Livanelioglu A, Soylu AR. Combined Effects of Mirror Therapy and Exercises on the Upper Extremities in Children with Unilateral Cerebral Palsy: A Randomized Controlled Trial. Dev Neurorehabil. 2020 May;23(4):253-264. doi: 10.1080/17518423.2019.1662853. Epub 2019 Sep 13. PMID 31514564
- [Background] Sirindhorn National Medical Rehabilitation Centre. Vojta therapy in childhood. Bangkok: Department of Medical Services, Ministry of Public Health; October 2556.
- [Background] Sung YH, Ha SY. The Vojta approach changes thicknesses of abdominal muscles and gait in children with spastic cerebral palsy: A randomized controlled trial, pilot study. Technol Health Care. 2020;28(3):293-301. doi: 10.3233/THC-191726. PMID 31658070
- [Background] Khiewcham P., Vongpipatana S., Wongphaet P., Thipsook K. Effect of Vojta Therapy on Gait of Children with Cerebral Palsy. J Thai Rehabil Med 2016; 26(3): 91-97
- [Background] Lim H, Kim T. Effects of vojta therapy on gait of children with spastic diplegia. J Phys Ther Sci. 2013 Dec;25(12):1605-8. doi: 10.1589/jpts.25.1605. Epub 2014 Jan 8. PMID 24409030
- [Background] Matic-Tec.de, S.R.| Therapie, Vojta. Available at: https://www.vojta.com/de/vojta-prinzip/vojtatherapie (Accessed: February 15, 2023).